CLINICAL TRIAL: NCT00162071
Title: "A Phase II Open-Label, Non-Randomized, Single-Center Trial to Determine the Optimal Myocardial Perfusion Image Acquisition Time Following BMS068645 Administration
Brief Title: A Phase II Optimization Study of BMS068645 and Sestamibi Planar Imaging
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decided not to continue with the development program
Sponsor: Forest Laboratories (Industry)
Responsible Party: Qi Zhu, MD Senior Medical Director, Lantheus Medical Imaging
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BMS068645-203
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Cardiovascular Disease; Ischemic Heart Disease
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Ischemia

INTERVENTIONS:
Drug: apadenoson

SUMMARY:
The primary purpose of this study is to determine the optimal time for myocardial perfusion imaging with Technetium Tc99m Sestamibi following the administration of BMS068645. The safety of BMS068645 will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Have known or suspected heart disease
* Have undergone a clinically indicated SPECT MPI study with adenosine in the last 24 hours to 14 days.
* Weigh between 88 and 250 lbs.

Exclusion Criteria:

* Allergic reaction to Technetium Tc99m Sestamibi or any of its components
* History of asthma or lung disease
* Ingestion of caffeinated substances within 12 hours prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-07; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Measurements of Technetium Tc99m Sestamibi activity will be obtained from various regions of the body at the end of the study to determine optimal imaging times.

SECONDARY OUTCOMES:
A comparison of adverse events will be conducted at the end of the study to assess safety.

CONTACTS AND LOCATIONS:
Overall Officials: E Gordon DePuey, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- Local Institution, New York, New York, United States